CLINICAL TRIAL: NCT04232800
Title: Riboflavin for Glutamate Reduction in Alcohol Withdrawal
Acronym: RGRAW
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Andrew Hughes, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RGRAW
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Alcohol Withdrawal; Nutrition Disorders; Alcohol Use Disorder
Keywords: Glutamate; Riboflavin
MeSH Terms: conditions — Nutrition Disorders; Alcoholism | interventions — Riboflavin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either riboflavin or an identical inert placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment and placebo capsules will be identical, and will be identified with each participants unique randomization number provided by the VA pharmacy. This will ensure blinding until study completion. Neither participants nor any study or treatment team members will know the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Riboflavin (Experimental): Participants in this group will receive 100mg riboflavin TID during study participation.
  Interventions: Drug: Riboflavin
- Placebo (Placebo Comparator): Participants in this group will receive inert placebo capsules TID during study participation.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Riboflavin — The intervention will consist of 100mg riboflavin (vitamin B2) given in three time daily dosing.
  Other Names: Vitamin B2
  Arms: Riboflavin
Other: Placebo — An inert, standard placebo in identical capsules to primary intervention.
  Arms: Placebo

SUMMARY:
This RCT intends to investigate the use of oral Riboflavin (Vitamin B2) for reduction of blood glutamate levels in the setting of acute alcohol withdrawal. Participants will be patients admitted to an inpatient hospital unit diagnosed with acute alcohol withdrawal. In addition to receiving care as usual, they will be randomized to receive either 100mg TID riboflavin or an identically dosed placebo. The primary outcome measure will be blood glutamate levels. Secondary outcomes will include measures of alcohol withdrawal and alcohol craving. The investigators hypothesize that those in the riboflavin group will have lower blood levels of glutamate, as well as decreased symptoms of alcohol withdrawal.

DETAILED DESCRIPTION:
General Investigational Plan

Hypotheses:

1. Aim 1: Measure the impact of daily oral riboflavin supplementation on blood Glu levels.

   Hypothesis 1: Patients receiving riboflavin will have significant reductions in blood Glu levels, as compared to placebo.
2. Aim 2: Observe the impact of oral riboflavin on CIWA-AR scale scoring. Hypothesis 2: Riboflavin will significantly reduce the active group's CIWA-AR scores, and will result in fewer symptom triggered benzodiazepine doses, as compared to placebo.

Plan: The proposed study would apply a recently identified method using vitamin B2 (riboflavin) to reduce excess brain Glu activity in veterans in acute alcohol withdrawal. This method of "glutamate scavenging", was identified in a 2018 as a way to reduce glutamate associated brain damage which typically occurs after stroke. When tested in human patients immediately following stroke, the intervention demonstrated efficacy through better structural and functional outcomes when compared to placebo. Improvements persisted at 3 months after the initial stroke, and were not associated with any known side effects. Administration of riboflavin quickly decreases Glu levels in both the blood and brain, as measured using chromatography and Magnetic Resonance Imaging (MRI), respectively. As riboflavin's Glu reducing properties have just been discovered, this method has only been applied to the treatment of stroke, and has yet to be studied outside of the field of neurology. Further, oral riboflavin has not been investigated as a method of glutamate reduction. The hyperglutamatergic state in patients with alcohol withdrawal provides one opportunity for such an investigation, one that may lead to future studies improving treatments of alcohol withdrawal. Chronic, as well as acute alcohol users have both elevated extracellular glutamate as well as changes to glutamate receptors and transporters. These changes appear play a role in the rewarding effects of alcohol, and contribute to the symptoms of withdrawal. A positive correlation exists between CSF levels of glutamate and the severity of alcohol dependence, and patients in acute withdrawal have measurably increased levels of glutamate in their peripheral blood. During early withdrawal, elevated glutamate levels have been observed in the hippocampus and anterior cingulate cortex, returning to normal 3 days after symptom resolution. Given this information, riboflavin may provide a safe, effective, and affordable intervention to normalize the hyperglutamatergic state associated with alcohol withdrawal. The proposed study would investigate this hypothesis in patients admitted to the inpatient psychiatry unit in acute alcohol withdrawal.

Methods: Participants would be recruited on the inpatient psychiatry unit as they were admitted. The primary teams/on call residents would be asked to page a study member if a patient was admitted on the standard protocol for alcohol withdrawal: the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar). The study coordinator would consent the patient, and they would be randomized to either the placebo or riboflavin group. They would then receive TID oral dosing of either 100mg riboflavin or placebo, in addition to treatment as usual. The primary outcome would be daily blood glutamate levels, obtained with the normal morning labs. Secondary outcomes would CIWA scores, number of symptom-triggered benzodiazepines given, anxiety, and alcohol craving scores (using standardized measures).

ELIGIBILITY:
Inclusion Criteria:

* Adult veterans ages 18-65
* Admitted to the inpatient psychiatric unit at the Portland VA
* Determine by admitting physician to be currently in or at risk of alcohol withdrawal during admission
* Placed on the CIWA-AR protocol
* Willing to provide informed consent/HIPAA authorization and accept randomization
* Willing to ingest three capsules/day
* Willing to provide daily blood samples H) Fluent in English

Exclusion Criteria:

* Known allergy to ingredients of riboflavin, capsules, or placebo ingredients
* Taking any medication acting primarily on Glu receptors (e.g. memantine) or GABA receptors (benzodiazepines) at baseline
* Unable to swallow capsules
* Actively in withdrawal from substances other than alcohol
* Unable to provide full informed consent/HIPAA authorization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-08-25 (Estimated); Study Completion 2022-10-25 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood glutamate level at baseline | Will occur on the day of enrollment in the study
  measured using high performance liquid chromatography (HPLC)
Peripheral blood glutamate level, day 2 | Will occur on day 2 of the study
  measured using high performance liquid chromatography (HPLC)
Peripheral blood glutamate level, day 4 | Will occur on day 4 of the study
  measured using high performance liquid chromatography (HPLC)
Peripheral blood glutamate level, day 6 | Will occur on day 6 of the study
  measured using high performance liquid chromatography (HPLC)
Peripheral blood glutamate level, day 8 | Will occur on day 8 of the study
  measured using high performance liquid chromatography (HPLC)
Peripheral blood glutamate level, day 10 | Will occur on day 10 of the study
  measured using high performance liquid chromatography (HPLC)

SECONDARY OUTCOMES:
Baseline Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale scores | Will occur on the day of enrollment in the study
  The CIWA-Ar scale is a measure used in standard of care treatment of alcohol withdrawal. It assesses severity of symptoms, and can be used to determine the need for supportive therapy (e.g. benzodiazepines).It will be collected as standard of care, and will be analyzed as a secondary outcome measure.Scores range from 0-67, with a higher number indicating increased symptoms of alcohol withdrawal.
Day 2: Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale scores | Will occur on the day 2 after randomization (if participant has not yet discharged from the hospital)
  The CIWA-Ar scale is a measure used in standard of care treatment of alcohol withdrawal. It assesses severity of symptoms, and can be used to determine the need for supportive therapy (e.g. benzodiazepines).It will be collected as standard of care, and will be analyzed as a secondary outcome measure.Scores range from 0-67, with a higher number indicating increased symptoms of alcohol withdrawal.
Day 3: Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale scores | Will occur on the day 3 after randomization (if participant has not yet discharged from the hospital)
  The CIWA-Ar scale is a measure used in standard of care treatment of alcohol withdrawal. It assesses severity of symptoms, and can be used to determine the need for supportive therapy (e.g. benzodiazepines).It will be collected as standard of care, and will be analyzed as a secondary outcome measure.Scores range from 0-67, with a higher number indicating increased symptoms of alcohol withdrawal.
Day 4: Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale scores | Will occur on the day 4 after randomization (if participant has not yet discharged from the hospital)
  The CIWA-Ar scale is a measure used in standard of care treatment of alcohol withdrawal. It assesses severity of symptoms, and can be used to determine the need for supportive therapy (e.g. benzodiazepines).It will be collected as standard of care, and will be analyzed as a secondary outcome measure.Scores range from 0-67, with a higher number indicating increased symptoms of alcohol withdrawal.
Day 5: Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale scores | Will occur on the day 5 after randomization (if participant has not yet discharged from the hospital)
  The CIWA-Ar scale is a measure used in standard of care treatment of alcohol withdrawal. It assesses severity of symptoms, and can be used to determine the need for supportive therapy (e.g. benzodiazepines).It will be collected as standard of care, and will be analyzed as a secondary outcome measure.Scores range from 0-67, with a higher number indicating increased symptoms of alcohol withdrawal.
Day 6: Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale scores | Will occur on the day 6 after randomization (if participant has not yet discharged from the hospital)
  The CIWA-Ar scale is a measure used in standard of care treatment of alcohol withdrawal. It assesses severity of symptoms, and can be used to determine the need for supportive therapy (e.g. benzodiazepines).It will be collected as standard of care, and will be analyzed as a secondary outcome measure.Scores range from 0-67, with a higher number indicating increased symptoms of alcohol withdrawal.
Day 7: Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale scores | Will occur on the day 7 after randomization (if participant has not yet discharged from the hospital)
  The CIWA-Ar scale is a measure used in standard of care treatment of alcohol withdrawal. It assesses severity of symptoms, and can be used to determine the need for supportive therapy (e.g. benzodiazepines).It will be collected as standard of care, and will be analyzed as a secondary outcome measure.Scores range from 0-67, with a higher number indicating increased symptoms of alcohol withdrawal.
Day 8: Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale scores | Will occur on the day 8 after randomization (if participant has not yet discharged from the hospital)
  The CIWA-Ar scale is a measure used in standard of care treatment of alcohol withdrawal. It assesses severity of symptoms, and can be used to determine the need for supportive therapy (e.g. benzodiazepines).It will be collected as standard of care, and will be analyzed as a secondary outcome measure.Scores range from 0-67, with a higher number indicating increased symptoms of alcohol withdrawal.
Day 9: Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale scores | Will occur on the day 9 after randomization (if participant has not yet discharged from the hospital)
  The CIWA-Ar scale is a measure used in standard of care treatment of alcohol withdrawal. It assesses severity of symptoms, and can be used to determine the need for supportive therapy (e.g. benzodiazepines).It will be collected as standard of care, and will be analyzed as a secondary outcome measure.Scores range from 0-67, with a higher number indicating increased symptoms of alcohol withdrawal.
Day 10: Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale scores | Will occur on the day 10 after randomization (if participant has not yet discharged from the hospital)
  The CIWA-Ar scale is a measure used in standard of care treatment of alcohol withdrawal. It assesses severity of symptoms, and can be used to determine the need for supportive therapy (e.g. benzodiazepines).It will be collected as standard of care, and will be analyzed as a secondary outcome measure.Scores range from 0-67, with a higher number indicating increased symptoms of alcohol withdrawal.
Baseline: # of Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale triggered benzodiazepine administration | Will occur on the day of enrollment in the study
  As part of standard of care for acute alcohol withdrawal, patients are administered benzodiazepines for symptoms if a clinician-determined threshold is met. That is, patients who are more symptomatic (higher CIWA-Ar) scores, receive more benzodiazepines. This data is collected as standard of care, but will be used as a secondary outcome for this study.
Day 2: # of Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale triggered benzodiazepine administration | Will occur on the day 2 after randomization (if participant has not yet discharged from the hospital)
  As part of standard of care for acute alcohol withdrawal, patients are administered benzodiazepines for symptoms if a clinician-determined threshold is met. That is, patients who are more symptomatic (higher CIWA-Ar) scores, receive more benzodiazepines. This data is collected as standard of care, but will be used as a secondary outcome for this study.
Day 3: # of Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale triggered benzodiazepine administration | Will occur on the day 3 after randomization (if participant has not yet discharged from the hospital)
  As part of standard of care for acute alcohol withdrawal, patients are administered benzodiazepines for symptoms if a clinician-determined threshold is met. That is, patients who are more symptomatic (higher CIWA-Ar) scores, receive more benzodiazepines. This data is collected as standard of care, but will be used as a secondary outcome for this study.
Day 4: # of Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale triggered benzodiazepine administration | Will occur on the day 4 after randomization (if participant has not yet discharged from the hospital)
  As part of standard of care for acute alcohol withdrawal, patients are administered benzodiazepines for symptoms if a clinician-determined threshold is met. That is, patients who are more symptomatic (higher CIWA-Ar) scores, receive more benzodiazepines. This data is collected as standard of care, but will be used as a secondary outcome for this study.
Day 5: # of Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale triggered benzodiazepine administration | Will occur on the day 5 after randomization (if participant has not yet discharged from the hospital)
  As part of standard of care for acute alcohol withdrawal, patients are administered benzodiazepines for symptoms if a clinician-determined threshold is met. That is, patients who are more symptomatic (higher CIWA-Ar) scores, receive more benzodiazepines. This data is collected as standard of care, but will be used as a secondary outcome for this study.
Day 6: # of Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale triggered benzodiazepine administration | Will occur on the day 6 after randomization (if participant has not yet discharged from the hospital)
  As part of standard of care for acute alcohol withdrawal, patients are administered benzodiazepines for symptoms if a clinician-determined threshold is met. That is, patients who are more symptomatic (higher CIWA-Ar) scores, receive more benzodiazepines. This data is collected as standard of care, but will be used as a secondary outcome for this study.
Day 7: # of Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale triggered benzodiazepine administration | Will occur on the day 7 after randomization (if participant has not yet discharged from the hospital)
  As part of standard of care for acute alcohol withdrawal, patients are administered benzodiazepines for symptoms if a clinician-determined threshold is met. That is, patients who are more symptomatic (higher CIWA-Ar) scores, receive more benzodiazepines. This data is collected as standard of care, but will be used as a secondary outcome for this study.
Day 8: # of Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale triggered benzodiazepine administration | Will occur on the day 8 after randomization (if participant has not yet discharged from the hospital)
  As part of standard of care for acute alcohol withdrawal, patients are administered benzodiazepines for symptoms if a clinician-determined threshold is met. That is, patients who are more symptomatic (higher CIWA-Ar) scores, receive more benzodiazepines. This data is collected as standard of care, but will be used as a secondary outcome for this study.
Day 9: # of Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale triggered benzodiazepine administration | Will occur on the day 9 after randomization (if participant has not yet discharged from the hospital)
  As part of standard of care for acute alcohol withdrawal, patients are administered benzodiazepines for symptoms if a clinician-determined threshold is met. That is, patients who are more symptomatic (higher CIWA-Ar) scores, receive more benzodiazepines. This data is collected as standard of care, but will be used as a secondary outcome for this study.
Day 10: # of Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale triggered benzodiazepine administration | Will occur on the day 10 after randomization (if participant has not yet discharged from the hospital)
  As part of standard of care for acute alcohol withdrawal, patients are administered benzodiazepines for symptoms if a clinician-determined threshold is met. That is, patients who are more symptomatic (higher CIWA-Ar) scores, receive more benzodiazepines. This data is collected as standard of care, but will be used as a secondary outcome for this study.
Baseline: Generalized Anxiety Disorder - 7 (GAD7) scale | Will occur on the day of enrollment in the study
  A standardized measure of anxiety over the previous 2 weeks. Scores range from 0-21, with a higher score indicating more symptoms of anxiety.
Day 2: Generalized Anxiety Disorder - 7 (GAD7) scale | Will occur on the day 2 after randomization (if participant has not yet discharged from the hospital)
  A standardized measure of anxiety over the previous 2 weeks. Scores range from 0-21, with a higher score indicating more symptoms of anxiety.
Day 3: Generalized Anxiety Disorder - 7 (GAD7) scale | Will occur on the day 3 after randomization (if participant has not yet discharged from the hospital)
  A standardized measure of anxiety over the previous 2 weeks. Scores range from 0-21, with a higher score indicating more symptoms of anxiety.
Day 4: Generalized Anxiety Disorder - 7 (GAD7) scale | Will occur on the day 4 after randomization (if participant has not yet discharged from the hospital)
  A standardized measure of anxiety over the previous 2 weeks. Scores range from 0-21, with a higher score indicating more symptoms of anxiety.
Day 5: Generalized Anxiety Disorder - 7 (GAD7) scale | Will occur on the day 5 after randomization (if participant has not yet discharged from the hospital)
  A standardized measure of anxiety over the previous 2 weeks. Scores range from 0-21, with a higher score indicating more symptoms of anxiety.
Day 6: Generalized Anxiety Disorder - 7 (GAD7) scale | Will occur on the day 6 after randomization (if participant has not yet discharged from the hospital)
  A standardized measure of anxiety over the previous 2 weeks. Scores range from 0-21, with a higher score indicating more symptoms of anxiety.
Day 7: Generalized Anxiety Disorder - 7 (GAD7) scale | Will occur on the day 7 after randomization (if participant has not yet discharged from the hospital)
  A standardized measure of anxiety over the previous 2 weeks. Scores range from 0-21, with a higher score indicating more symptoms of anxiety.
Day 8: Generalized Anxiety Disorder - 7 (GAD7) scale | Will occur on the day 8 after randomization (if participant has not yet discharged from the hospital)
  A standardized measure of anxiety over the previous 2 weeks. Scores range from 0-21, with a higher score indicating more symptoms of anxiety.
Day 9: Generalized Anxiety Disorder - 7 (GAD7) scale | Will occur on the day 9 after randomization (if participant has not yet discharged from the hospital)
  A standardized measure of anxiety over the previous 2 weeks. Scores range from 0-21, with a higher score indicating more symptoms of anxiety.
Day 10: Generalized Anxiety Disorder - 7 (GAD7) scale | Will occur on the day 10 after randomization (if participant has not yet discharged from the hospital)
  A standardized measure of anxiety over the previous 2 weeks. Scores range from 0-21, with a higher score indicating more symptoms of anxiety.
Baseline: The Alcohol Craving Questionnaire-Revised (ACQ-R) | Will occur on the day of enrollment in the study
  A brief, reliable, and validated measure of alcohol craving. Scores range from 1-7 with higher scores indicating stronger alcohol cravings
Day 2: The Alcohol Craving Questionnaire-Revised (ACQ-R) | Will occur on the day 2 after randomization (if participant has not yet discharged from the hospital)
  A brief, reliable, and validated measure of alcohol craving. Scores range from 1-7 with higher scores indicating stronger alcohol cravings
Day 3: The Alcohol Craving Questionnaire-Revised (ACQ-R) | Will occur on the day 3 after randomization (if participant has not yet discharged from the hospital)
  A brief, reliable, and validated measure of alcohol craving. Scores range from 1-7 with higher scores indicating stronger alcohol cravings
Day 4: The Alcohol Craving Questionnaire-Revised (ACQ-R) | Will occur on the day 4 after randomization (if participant has not yet discharged from the hospital)
  A brief, reliable, and validated measure of alcohol craving. Scores range from 1-7 with higher scores indicating stronger alcohol cravings
Day 5: The Alcohol Craving Questionnaire-Revised (ACQ-R) | Will occur on the day 5 after randomization (if participant has not yet discharged from the hospital)
  A brief, reliable, and validated measure of alcohol craving. Scores range from 1-7 with higher scores indicating stronger alcohol cravings
Day 6: The Alcohol Craving Questionnaire-Revised (ACQ-R) | Will occur on the day 6 after randomization (if participant has not yet discharged from the hospital)
  A brief, reliable, and validated measure of alcohol craving. Scores range from 1-7 with higher scores indicating stronger alcohol cravings
Day 7: The Alcohol Craving Questionnaire-Revised (ACQ-R) | Will occur on the day 7 after randomization (if participant has not yet discharged from the hospital)
  A brief, reliable, and validated measure of alcohol craving. Scores range from 1-7 with higher scores indicating stronger alcohol cravings
Day 8: The Alcohol Craving Questionnaire-Revised (ACQ-R) | Will occur on the day 8 after randomization (if participant has not yet discharged from the hospital)
  A brief, reliable, and validated measure of alcohol craving. Scores range from 1-7 with higher scores indicating stronger alcohol cravings
Day 9: The Alcohol Craving Questionnaire-Revised (ACQ-R) | Will occur on the day 9 after randomization (if participant has not yet discharged from the hospital)
  A brief, reliable, and validated measure of alcohol craving. Scores range from 1-7 with higher scores indicating stronger alcohol cravings
Day 10: The Alcohol Craving Questionnaire-Revised (ACQ-R) | Will occur on the day 10 after randomization (if participant has not yet discharged from the hospital)
  A brief, reliable, and validated measure of alcohol craving. Scores range from 1-7 with higher scores indicating stronger alcohol cravings
Baseline: The Daily Assessment of Symptoms -Anxiety (DAS-A) | Will occur on the day of enrollment in the study
  A reliable and valid measure of anxiety which has been shown to detect reduction of anxiety symptoms within 24 hours. Scores range from 0-80, with a higher score indicating more symptoms of anxiety
Day 2: The Daily Assessment of Symptoms -Anxiety (DAS-A) | Will occur on the day 2 after randomization (if participant has not yet discharged from the hospital)
  A reliable and valid measure of anxiety which has been shown to detect reduction of anxiety symptoms within 24 hours. Scores range from 0-80, with a higher score indicating more symptoms of anxiety
Day 3: The Daily Assessment of Symptoms -Anxiety (DAS-A) | Will occur on the day 3 after randomization (if participant has not yet discharged from the hospital)
  A reliable and valid measure of anxiety which has been shown to detect reduction of anxiety symptoms within 24 hours. Scores range from 0-80, with a higher score indicating more symptoms of anxiety
Day 4: The Daily Assessment of Symptoms -Anxiety (DAS-A) | Will occur on the day 4 after randomization (if participant has not yet discharged from the hospital)
  A reliable and valid measure of anxiety which has been shown to detect reduction of anxiety symptoms within 24 hours. Scores range from 0-80, with a higher score indicating more symptoms of anxiety
Day 5: The Daily Assessment of Symptoms -Anxiety (DAS-A) | Will occur on the day 5 after randomization (if participant has not yet discharged from the hospital)
  A reliable and valid measure of anxiety which has been shown to detect reduction of anxiety symptoms within 24 hours. Scores range from 0-80, with a higher score indicating more symptoms of anxiety
Day 6: The Daily Assessment of Symptoms -Anxiety (DAS-A) | Will occur on the day 6 after randomization (if participant has not yet discharged from the hospital)
  A reliable and valid measure of anxiety which has been shown to detect reduction of anxiety symptoms within 24 hours. Scores range from 0-80, with a higher score indicating more symptoms of anxiety
Day 7: The Daily Assessment of Symptoms -Anxiety (DAS-A) | Will occur on the day 7 after randomization (if participant has not yet discharged from the hospital)
  A reliable and valid measure of anxiety which has been shown to detect reduction of anxiety symptoms within 24 hours. Scores range from 0-80, with a higher score indicating more symptoms of anxiety
Day 8: The Daily Assessment of Symptoms -Anxiety (DAS-A) | Will occur on the day 8 after randomization (if participant has not yet discharged from the hospital)
  A reliable and valid measure of anxiety which has been shown to detect reduction of anxiety symptoms within 24 hours. Scores range from 0-80, with a higher score indicating more symptoms of anxiety
Day 9: The Daily Assessment of Symptoms -Anxiety (DAS-A) | Will occur on the day 9 after randomization (if participant has not yet discharged from the hospital)
  A reliable and valid measure of anxiety which has been shown to detect reduction of anxiety symptoms within 24 hours. Scores range from 0-80, with a higher score indicating more symptoms of anxiety
Day 10: The Daily Assessment of Symptoms -Anxiety (DAS-A) | Will occur on the day 10 after randomization (if participant has not yet discharged from the hospital)
  A reliable and valid measure of anxiety which has been shown to detect reduction of anxiety symptoms within 24 hours. Scores range from 0-80, with a higher score indicating more symptoms of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Cornejo, MD, PhD, Principal Investigator — Oregon Health & Science University, Portland Veterans Health Administration

IPD SHARING:
Plan to Share IPD: No